CLINICAL TRIAL: NCT06882746
Title: A Phase I, Open-label, Non-randomised, Multi-center Dose Escalation Trial of BI 765049 Administered by Parenteral Route in Patients With Advanced, Unresectable, and/or Metastatic Colorectal Carcinoma (CRC), Gastric Carcinoma (GC), or Pancreatic Ductal Adenocarcinoma (PDAC) to Determine the MTD and the RP2D and to Determine the Dosing Regimen for Further Development of BI 765049
Brief Title: A Study to Test Different Doses of BI 765049 in People With Advanced Cancer of the Colon, Rectum, Stomach, or Pancreas
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1454-0015; 2024-519301-36-00 (EU CTIS Number); U1111-1316-8363 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-03-17; First posted 2025-03-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Carcinoma; Gastric Carcinoma; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Part 1 and part 2 run in parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Administration Regimen A) (Experimental)
  Interventions: Drug: BI 765049
- Part 2 (Administration Regimen B) (Experimental)
  Interventions: Drug: BI 765049

INTERVENTIONS:
Drug: BI 765049 — BI 765049

SUMMARY:
This study is open to adults with advanced cancer of the colon, rectum, stomach, or pancreas, that is the cancer cannot be removed by surgery or has spread. People can take part in this study if their previous treatment was not successful, or no other treatment exists.

The study aims to find the highest dose for the study medicine called BI 765049 that people with advanced cancer can tolerate. Another purpose is to find the most suitable dose and best way of administration of BI 765049 for further clinical development. BI 765049 may help the immune system fight cancer.

Participants receive BI 765049 at least once every 3 weeks. Participants may continue to get BI 765049 treatment as long as they benefit from treatment and can tolerate it.

During this time, participants regularly visit the study site. The study visits include several overnight stays at the hospital. At the visits, study doctors check participants' health, take necessary laboratory tests, and note any unwanted effects. Unwanted effects are any health problems that the doctors think were caused by the study medicine or treatment. To find the highest dose of BI 765049 that participants can tolerate, researchers look at the number of participants with certain severe health problems. These are severe health problems that happen within 1 week after the first treatment with the intended dose.

ELIGIBILITY:
Inclusion criteria:

* Signed and dated informed consent form (ICF)2/main ICF for all patients describing the study in accordance with International Council on Harmonisation Good Clinical Practice (ICH-GCP) and local legislation prior to any trial-specific procedures, sampling, or analyses.
* Patient must be ≥18 years of age and at least at the legal age of consent in countries where it is greater than 18 years at the time of signature on the ICFs (ICF1/screening ICF and ICF2/main ICF).
* In US: Patients with a histologically or cytologically confirmed diagnosis of colorectal carcinoma (CRC), gastric carcinoma (GC), or pancreatic ductal adenocarcinoma (PDAC).
* In Europe: Patients with a histologically or cytologically confirmed diagnosis of CRC.
* Patients with advanced, unresectable, and/or metastatic disease. Further inclusion criteria apply.

Exclusion criteria:

* Patient with a history of a major surgery within 28 days prior to first dose of BI 765049 (major according to the Investigator's and/or Medical Monitor's assessment).
* Previous or concomitant malignancies other than the one treated in this trial within the last 5 years except:

  * Effectively treated non-melanoma skin cancers
  * Effectively treated carcinoma in situ of the cervix
  * Effectively treated ductal carcinoma in situ
  * Other effectively treated malignancy that is considered cured by local treatment"
* Patient with known leptomeningeal disease or spinal cord compression due to disease.
* Patient requiring anticoagulant treatment which cannot be safely interrupted, if medically needed based on the opinion of the Investigator.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities (DLTs) in the maximum tolerated dose (MTD) evaluation period | up to 36 months

SECONDARY OUTCOMES:
Objective response (OR) | up to 36 months
  OR defined as the best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to response evaluation criteria in solid tumors (RECIST) 1.1 from the date of treatment start until the earliest date of disease progression, death, or last evaluable tumor assessment before start of subsequent anti-cancer therapy, or treatment discontinuation as assessed by investigator review
Occurrence of DLTs and adverse events during the entire treatment period | up to 36 months
Maximum measured concentration (Cmax) of BI 765049 after first administration | up to 4 days
Maximum measured concentration (Cmax) of BI 765049 after multiple administrations | up to 20 days
Area under the concentration-time curve of BI 765049 over a uniform dosing interval τ (AUCτ) after first administration | up to 4 days
Area under the concentration-time curve of BI 765049 over a uniform dosing interval τ (AUCτ) after multiple administrations | up to 20 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Valkyrie Clinical Trials, Los Angeles, California
  - Winship Cancer Institute, Atlanta, Georgia
  - Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com